CLINICAL TRIAL: NCT04970264
Title: A Observational RWS of YWBC on the Prognosis and Treatment
Brief Title: A Multicenter, Open and Observational Real World Study on the Prognosis and Treatment in Young Women With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YWBC-001
Record Dates: First submitted 2021-02-26; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: young women with breast cancer; gene mutation characteristics; prognosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Fresh tissue from surgery or puncture, or formalin-fixed paraffin-embedded (FFPE) sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, open and observational real world study. The main purpose of this study is to map the genomic variation map of young breast cancer patients in China, and to analyze the relationship between gene mutation and therapeutic effect of young breast cancer patients. The secondary purpose was to analyze the relationship between gene mutation and prognosis of young breast cancer patients.

We expect to enroll 2000 young breast cancer patients (≤35 years old). All patients were detected by targeted next generation sequencing （NGS）(600+ gene panel). Clinical diagnosis, treatment and prognosis information were collected. The Stratification factors mainly include stage, molecular type and treatment method.

DETAILED DESCRIPTION:
The study can only be formally carried out with the written approval of the ethics committee. We regularly submit annual research reports to the ethics committee. We will inform the ethics committee in writing when the study is discontinued and / or completed.

All patients were required to sign informed consent before entering the group. All updated versions of informed consent and written information will be provided to the subjects during the participant's participation.

In the experimental design stage, the statistical principle was used to make reasonable and effective arrangements for the relevant factors. Employ statistical experts to calculate the sample size and data statistics, and participate in the design process. Data collection and follow-up were conducted by specially assigned personnel, professional doctors were assigned to conduct data review regularly, and special data management personnel were provided. They will ensure the authenticity, reliability and security of data throughout the process.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed as breast cancer.
2. The age of diagnosis was 18-35 years old.
3. ECOG score was 0-2, and the expected survival time was more than 3 months.
4. No serious complications; no liver, kidney, hematopoiesis dysfunction.
5. Informed consent, and patients willing to long-term follow-up. -

Exclusion Criteria:

1. 4 weeks before the start of the study, the use of drugs other than the trial, or participate in another clinical study at the same time, or others with an impact on the results of this study.
2. Having a clear history of neurological or mental disorders (including epilepsy or dementia).
3. Patients have uncontrollable complications, including active infection, symptomatic congestive heart failure, unstable angina pectoris, arrhythmia, decompensated diabetes, uncontrollable hypertension or mental disorders.
4. Pregnant or lactating female patients.
5. HIV infected patients.
6. Patients with other tumors.
7. After comprehensive evaluation, the researchers believe that patients are not suitable for this study.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: We expect to enroll 2000 young breast cancer patients (18-35 years old). All patients were detected by targeted next generation sequencing （NGS）(600+ gene panel).
  Subgroups were stratified according to different stages, treatment methods and pathological types.
  The gene mutation characteristics, treatment sensitive genes and prognosis gene spectrum of different groups and subgroups were studied.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years
  The time from the first medication at the beginning of treatment to the first disease progression or death from any cause

SECONDARY OUTCOMES:
OS | 5 years
  time from randomization to death from any cause
ORR | 5 years
  After treatment, the percentage of patients whose tumor volume reduced to a predetermined value and could maintain the minimum time limit was evaluated, including complete remission (CR) + partial remission (PR)

OTHER OUTCOMES:
AEs | 5 years
  It refers to any adverse medical event during the clinical study. It is not necessarily a causal relationship with treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- TianJin Medical University Cancer Institute and Hospital, Tianjin, China